CLINICAL TRIAL: NCT00274248
Title: A Phase 1 Study of MLN518 Given in Combination With Standard Induction Chemotherapy for the Treatment of Patients With Newly Diagnosed Acute Myelogenous Leukemia
Brief Title: MLN518 in Combination With Standard Induction Chemo. for Treatment of Patients With Newly Diagnosed Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C03001
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tandutinib

INTERVENTIONS:
Drug: MLN518

SUMMARY:
This is a phase 1, open-label, multicenter study investigating the use of MLN518 in combination with standard chemotherapy to patients with newly diagnosed AML. Two dose levels of MLN518-200 mg and 400 mg given orally twice a day are planned for sequential evaluation in separate groups of patients. Patients assigned to the 400 mg dose level given orally twice a day of MLN518, will potentially have their dose of MLN518 adjusted on the basis of MLN518 plasma concentrations measured during the first 3 days of induction therapy. All patients will receive initial induction chemotherapy with cytarabine, 200 mg/m2/day by CIVI on Days 1 through 7, and with daunorubicin, 60 mg/m2/day by intravenous (IV) push (IV infusion if borderline cardiac function is detected) on Days 1 through 3 ("7+3"). An abbreviated cytarabine and daunorubicin regimen ("5+2") will also be used when the initial remission induction therapy fails to clear the bone marrow of blast cells (as typically detected on the Day 15 bone marrow) and a second attempt at remission induction is indicated. Patients who achieve a complete remission (CR) will receive consolidation therapy with HiDAC (standard or modified) in combination with continued MLN518 treatment. Patients remaining in continuous CR after completion of their last cycle of consolidation therapy will be permitted to continue treatment with single-agent MLN518 for 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, at least 18 years of age, with newly diagnosed (previously untreated) AML, regardless of the mutational status of FLT3 in their leukemic blasts.
* Unequivocal histologic diagnosis of AML (based on the World Health Organization [WHO] and/or FAB classifications), excluding acute promyelocytic leukemia. AML patients with a history of antecedent myelodysplasia (MDS) are eligible for treatment in this trial but must not have had prior cytotoxic therapy for MDS.
* No prior anti-neoplastic therapy for leukemia or MDS with the following exceptions:

  * emergency leukapheresis;
  * emergency treatment for hyperleukocytosis with hydroxyurea;
  * growth factor/cytokine support.
* Eastern Cooperative Oncology Group performance status of 0 to 3
* Pretreatment laboratory test values within the following limits no more than 7 days before enrollment:

  * total bilirubin equal or less then 1.5 x the upper limit of normal;
  * Alanine aminotransferase and aspartate aminotransferase equal or less then 2.5 x the ULN;
  * serum creatinine equal or less then 2.0 mg/dL.
* Male patients must use an appropriate method of barrier contraception during the study.
* Female patients must be postmenopausal, surgically sterilized, or willing to use reliable methods of birth control (ie, a hormonal contraceptive, an intrauterine device, diaphragm with spermicide, or abstinence) for the duration of the study.
* Ability to voluntarily provide written informed consent before the performance of any study related procedure not part of normal medical care.

Exclusion Criteria:

* An active malignancy other than AML (with the exception of basal and/or squamous cell skin cancers and curatively treated carcinoma of the cervix) at the time of study entry.
* Suspected or confirmed diagnosis of acute promyelocytic leukemia [t (15;17)(q22;q12)].
* Documented or suspected central nervous system (CNS) involvement with leukemia.
* Ongoing vomiting.
* Nausea of intensity greater than Grade 1 based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) categorization.
* Known gastrointestinal disease that could interfere with the oral absorption of MLN518.
* Severe CNS, pulmonary, renal, or hepatic disease not related to the patient's AML.
* A left ventricular ejection fraction < 40%.
* Myocardial infarction within 6 months of enrollment or New York Heart Association (NYHA) Class III or IV heart failure (see Appendix 3), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* QTc > 500 msec.
* Known or suspected infection with human immunodeficiency virus (HIV).
* Known active infection with hepatitis B or hepatitis C.
* Known or suspected primary muscular or neuromuscular disease (eg, muscular dystrophy, myasthenia gravis).
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Inability to provide written informed consent to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-03; Primary Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Dana Farber Cancer Institute, Boston, Massachusetts, United States